CLINICAL TRIAL: NCT00702689
Title: A Phase II Study of Imatinib Mesylate in Children and Adults With Sclerotic Skin Changes of Chronic Graft-Versus-Host Disease
Brief Title: Imatinib Mesylate to Treat Skin Changes in Patients With Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Cowen, M.D., Principal Investigator, National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080148; 08-AR-0148
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Sclerotic Graft Versus Host Disease; Imatinib Mesylate
Keywords: Skin Sclerosis; Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imatinib mesylate in patients with cGVHD (Experimental): Cohort 1 - Pts 1-8:Adults: 400mg imatinib mesylate daily; Children: 260mg/m^2 daily (400mg maximum), followed by dose de-escalation for adverse events.
  Cohort 2 - Pts 9-20:Adults - 100 mg oral dose daily (increase to 200 mg daily after 28 days if well tolerated). Children - 65 mg/m^2 oral dose daily (increase to 130 mg/m^2 daily after 28 days if well tolerated)
  Interventions: Drug: Gleevec, STI571(Imatinib Mesylate)

INTERVENTIONS:
Drug: Gleevec, STI571(Imatinib Mesylate) — Cohort 1 - Pts 1-8:Adults: 400mg imatinib mesylate daily; Children: 260mg/m^2 daily (400mg maximum), followed by dose de-escalation for adverse events.
  Cohort 2 - Pts 9-20:Adults - 100 mg oral dose daily (increase to 200 mg daily after 28 days if well tolerated). Children - 65 mg/m^2 oral dose daily (increase to 130 mg/m^2 daily after 28 days if well tolerated)
  Other Names: Gleevec; ST1571

SUMMARY:
Background:

Chronic graft-versus-host disease (GVHD) is a common complication of stem cell transplant, resulting from the donor's immune cells attacking the cells of the body of the recipient. One effect of GVHD is fibrosis (scarring) of the skin that can lead to impaired function, decreased quality of life and increased risk of death. This is known as sclerotic skin changes of GVHD, or sclerodermatous graft versus host disease (ScGVHD).

Imatinib mesylate (Gleevec) is a drug that has been approved by the Food and Drug Administration to treat cancer in humans and fibrosing conditions in animals.

Objectives:

To see if imatinib mesylate can improve ScGVHD and evaluate its effect on other GVHD symptoms

To assess the side effects of imatinib mesylate in patients with GVHD

To evaluate blood, body fluids and tissue samples in patients to try to better understand the biology of ScGVHD

Eligibility:

Patients 4 years of age and older with ScGVHD

Design:

Initial treatment: Participants take imatinib mesylate tablets once a day for up to 6 months, as long as their GVHD does not get worse and they do not develop unacceptable side effects of the drug.

Evaluations: Participants are evaluated at 1, 3 and 6 months at the National Institutes of Health (NIH) Clinical Center with procedures that may include the following:

Medical history and physical examination

Blood and urine tests

Lung function test

Skin biopsy

Magnetic resonance imaging (MRI) scan

Specialty consultations (e.g., physical or rehabilitative therapy, dentist, eye doctor, dermatologist)

Electrocardiogram (EKG)

Echocardiogram (ultrasound test of the heart)

Muga scan (nuclear medicine test of the heart)

Quality-of-life questionnaires

Apheresis (procedure for collecting quantities of white blood cells)

Office visits with local physician once a week for 1 month, then once every 2 weeks for 5 months

Followup visits at National Institutes of Health (NIH) every 6 months for 1 year

Continuing treatment: Patients who improve continue to receive imatinib mesylate for up to 6 months after their best response and are followed for up to 2 years. Patients who continue to respond or who become worse after stopping treatment may receive additional treatment for up to 2 years.

DETAILED DESCRIPTION:
Background:

Chronic graft versus host disease (cGVHD) is a major complication of allogeneic stem cell transplant (alloHSCT). The sclerotic skin manifestations of chronic cutaneous GVHD (ScGVHD) can lead to significant functional impairment and no satisfactory therapy exists to adequately treat this form of cGVHD.

Imatinib mesylate (Gleevec) is a small molecule tyrosine kinase inhibitor with potent activity against platelet derived growth factor receptor (PDGFR) signaling, a key cytokine pathway which has been implicated in fibrotic disease in general, and in extensive cGVHD in particular.

We hypothesize that treatment with imatinib mesylate will reduce the sclerotic manifestations of cGVHD as assessed by quantitative range of motion assessment of an affected joint.

Objectives:

Primary Objective:

To investigate whether imatinib mesylate results in clinical improvement in skin fibrosis in children and adults with ScGVHD using range of motion assessment of affected joints.

To determine if imatinib mesylate 200 mg daily is tolerated by patients with cGVHD.

Secondary Objectives:

To assess toxicity associated with imatinib mesylate in patients with cGVHD.

To establish outcome criteria for the evaluation of ScGVHD using multi-modality objective and subjective assessments, including magnetic resonance imaging, skin scoring, and patient self-reported measures.

To evaluate biomarkers of disease activity and correlative response measures to treatment with imatinib mesylate.

To assess quality of life and functional measures of disease activity and to evaluate changes through the course of therapy.

To evaluate the response of other organ manifestations affected by cGVHD to treatment with imatinib mesylate.

To evaluate steady-state pharmacokinetics of imatinib mesylate in the cGVHD patient population.

Eligibility:

Patients age 4 years of age or older with the diagnosis of ScGVHD.

Design:

This is an open-label, pilot study of imatinib mesylate.

Treatment cycles are 28-day cycles with no rest period between cycles.

A target of 10 evaluable patients will be enrolled on this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Sclerodermatous graft versus host disease (ScGVHD) manifesting after at least 100 days following allogeneic hematopoietic stem cell transplantation is considered diagnostic for chronic graft versus host disease (cGVHD) according to National Institutes of Health (NIH) cGVHD Consensus Statement diagnostic criteria.

This diagnosis can be made clinically or by histopathology. The diagnosis must be confirmed by the principal investigator (PI), or lead associate investigator (LAI).

Skin biopsies will be reviewed by the National Cancer Institute (NCI) Laboratory of Pathology to confirm the diagnosis of ScGVHD.

* Patients must have measurable limitation in range of motion, defined as ScGVHD with or without fasciitis, restricting range of motion (ROM) of at least one joint with a minimum deficit of 25 percent.
* Prior therapy: Patients must have cGVHD refractory to at least one treatment regimen for cGVHD.

One prior regimen must have included systemic corticosteroids at the equivalent prednisone dosing of 1mg/kg/day times 14 days.

Patients in whom calcineurin inhibitors or corticosteroids are medically contraindicated may also be eligible for enrollment.

Patients who have had stabilization of disease on calcineurin inhibitors or steroids, but in whom these medications cannot be tapered without disease flare are also eligible.

Patient must be on stable or tapering immunosuppressive regimen for at least one month.

* Age: 4 years of age or older at the time of enrollment. Lower age limit set by lower established age limit norms of ROM scores for measurement criteria.
* Life expectancy of greater than 6 months.
* Karnofsky greater than or equal to 60 percent.
* Patients must be platelet transfusion and growth factor independent at the time of study entry.

Patients must have adequate organ and marrow function as defined below. Patients with Gilbert syndrome are excluded from the requirement of a normal bilirubin.

(Gilbert syndrome is found in 3-10 percent of the general population, and is characterized by mild, chronic unconjugated hyperbilirubinemia in the absence of liver disease or overt hemolysis).

* absolute neutrophil count greater than or equal to 1,000/mcL
* platelets greater than or equal to 50,000/mcL
* total bilirubin less than 3 times upper limit of normal
* aspartate aminotransferase (AST)serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)serum glutamic pyruvic transaminase (SGPT) less than 5 times upper limit of normal
* creatinine age-adjusted within normal limits

OR

* creatinine clearance greater than 20mL/min/1.73 m^2 for adults and pediatric patients with body surface area (BSA) greater than 0.97 m^2 with creatinine levels above institutional normals and greater than or equal to 40 mL/min 1.73 m^2 for pediatric patients with BSA less than 0.97 m^2.
* Age less than 5 years old Maximum Serum Creatinine 0.8 mg/dL
* Age 5 or less than 10 years old Maximum Serum Creatinine 1.0 mg/dL
* Age 10 or less than 15 years old Maximum Serum Creatinine 1.2 mg/dL
* Age 15 years old or greater Maximum Serum Creatinine 1.5 mg/dL
* Normal cardiac function for age as determined by echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) (normal left ventricular (LV) function as measured by ejection fraction or shortening fraction).
* The effects of imatinib mesylate on the developing human fetus at the recommended therapeutic dose are unknown.

For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for six months following completion of therapy.

Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

* Ability to understand and the willingness to sign a written informed consent document.

All patients or their legal guardian (for patients less than 18 years old) must sign an institutional review board (IRB) approved document of informed consent (chronic graft versus host disease (cGVHD) natural history or any National Cancer Institute (NCI) protocol allowing for screening procedures) prior to performing studies to determine patient eligibility.

After confirmation of patient eligibility all patients or their legal guardian must sign the protocol-specific informed consent.

Pediatric patients will be included in age appropriate discussions and age appropriate assent will be obtained in accordance with National Institutes of Health (NIH) guidelines.

* Durable Power of Attorney (DPA): All patients 18 years of age at the time of enrollment will be offered the opportunity to assign DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy, radiotherapy, or immunotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents, including extracorporeal photopheresis.

Patients may not have received monoclonal antibody therapy within 6 weeks.

* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imatinib mesylate.
* Patients receiving any of the following medications or substances that are inhibitors or inducers of P450 3A4 are ineligible.

Use of the following medications must be discontinued at least two weeks prior to starting therapy:

* Alfuzosin
* Aprepitant
* Carbamazepine
* Clarithromycin
* Eletriptan
* Erythromycin
* Pimozide
* St John's Wort
* Warfarin
* A list of medications and substances known or with the potential to interact with the P450 3A4 isoenzyme is provided in Section 8.

Imatinib mesylate is likely to increase the blood level of drugs that are substrates of CYP2C9, CYP2D6 and CYP3A4/5.

Close monitoring is warranted when using agents metabolized by these enzymes. Grapefruit juice should not be consumed while on therapy.

* Prior treatment with imatinib mesylate or other tyrosine kinase inhibitor after the date of transplant.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary, hepatic, or other organ dysfunction, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the patient's ability to tolerate protocol therapy.
* Pregnant women are excluded from this study because imatinib mesylate is an agent with the potential for teratogenic or abortifacient effects.

Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with imatinib mesylate, breastfeeding should be discontinued if the mother is treated with imatinib mesylate.

* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with imatinib mesylate and the possibility of associated severe immunosuppression.
* Patients with active hepatitis C or hepatitis B infection as defined by seropositivity for hepatitis C or hepatitis B (HepBSAg) and elevated transaminases, as GVHD manifestations involving the liver will be indistinguishable and drug-toxicity uninterpretable.
* Persistent malignancy, requiring ongoing therapy.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12-15 (Actual); Primary Completion 2011-05-18 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Cowen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baird K, Comis LE, Joe GO, Steinberg SM, Hakim FT, Rose JJ, Mitchell SA, Pavletic SZ, Figg WD, Yao L, Flanders KC, Takebe N, Sarantopoulos S, Booher S, Cowen EW. Imatinib mesylate for the treatment of steroid-refractory sclerotic-type cutaneous chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2015 Jun;21(6):1083-90. doi: 10.1016/j.bbmt.2015.03.006. Epub 2015 Mar 12. PMID 25771402
- [Derived] Rosenthal EA, Ho PS, Joe GO, Mitchell SA, Booher S, Pavletic SZ, Baird K, Cowen EW, Comis LE. Motor ability, function, and health-related quality of life as correlates of symptom burden in patients with sclerotic chronic graft-versus-host disease receiving imatinib mesylate. Support Care Cancer. 2020 Aug;28(8):3679-3689. doi: 10.1007/s00520-019-05207-z. Epub 2019 Dec 6. PMID 31811481
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0148.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Started | 20
Completed | 14
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Recurrent malignancy | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.59 (17.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Chronic Graft Versus Host Disease (cGVHD) category [Number; unit: percentage of participants]
  Overlap | 5
  Classic | 95
  Late acute | 0
Chronic Graft Versus Host Disease presentation [Number; unit: Percentage of participants]
  De novo | 30
  Quiescent | 20
  Progressive | 50
Global National Institutes of Health Graft Versus Host Disease (GVHD) score [Number; unit: Percentage of participants]
  Mild (1) | 0
  Moderate (2) | 0
  Severe (3) | 100
Donor Source [Number; unit: Percentage of participants]
  Bone marrow | 10
  Peripheral blood | 90
  Cord | 0
Donor Match (6/6) [Number; unit: Percentage of participants] | 90
Months from Chronic Graft Versus Host Disease (cGVHD) diagnosis [Median (Full Range); unit: Months] | 39.85 [4.8 to 112]
Months from transplant [Median (Full Range); unit: Months] | 55.4 [12.7 to 121]
Concomitant Immunosuppressive Medication (ISM) [Count of Participants; unit: Participants] — Pred:prednisone; tacro:tacrolimus; MPred:methylprednisolone; MTX:methotrexate; siro:sirolimus; and MMF:mycophenolate mofetil
  Participants
    Pred/tacro | 2
    Pred | 1
    MPred/MTX | 1
    Pred/siro | 2
    Pred/siro/tacro | 1
    MPred/tacro/siro/MMF | 1
    Pred/siro/MMF | 2
    Tacro | 1
    Pred/tacro/siro | 1
    Tacro/MMF | 3
    Pred/MMF | 1
    Siro/MMF | 1
    MPred/tacro/MMF | 1
    Siro | 1
    None | 1
Assessable Joints at Baseline [Number; unit: joints] — *Patient 13 started with 3 measurable joints at enrollment on study. Patient experienced an episode of acute shoulder pain while on study, and evaluation revealed avascular necrosis of that shoulder. Therefore, only 2 joints were used in the final analysis.
  joints
    Patient 1 | 3
    Patient 2 | 3
    Patient 3 | 2
    Patient 4 | 3
    Patient 5 | 3
    Patient 6 | 3
    Patient 7 | 3
    Patient 8 | 3
    Patient 9 | 3
    Patient 10 | 3
    Patient 11 | 3
    Patient 12 | 3
    *Patient 13 | 3
    Patient 14 | 3
    Patient 15 | 3
    Patient 16 | 1
    Patient 17 | 3
    Patient 18 | 3
    Patient 19 | 3
    Patient 20 | 3
Average National Institutes of Health Chronic Graft Versus Host Disease (cGVHD) Score at Baseline [Number; unit: scores on a scale] — The scores are the average scores for each patient based on the sum of individual organ involvement (0-3) for 7 organs (males) and 8 organs (females) divided by 7 or 8, respectively. This is demographic data and no measure of dispersion was performed. An organ score of zero is none, and 3 is severely affected.
  scores on a scale
    Patient 1 | 1.28
    Patient 2 | 1.14
    Patient 3 | .75
    Patient 4 | 1.0
    Patient 5 | 1.48
    Patient 6 | 1.86
    Patient 7 | 1.90
    Patient 8 | 1.57
    Patient 9 | 1.71
    Patient 10 | 1.43
    Patient 11 | 1.75
    Patient 12 | 1.43
    Patient 13 | 1.38
    Patient 14 | 1.29
    Patient 15 | 1.43
    Patient 16 | .86
    Patient 17 | 1.13
    Patient 18 | 1.57
    Patient 19 | 1.14
    Patient 20 | 2.00
Measure of Number of Organs with Graft Versus Host Disease (GVHD) [Number; unit: affected organs]
  Patient 1 | 5
  Patient 2 | 4
  Patient 3 | 3
  Patient 4 | 4
  Patient 5 | 6
  Patient 6 | 7
  Patient 7 | 7
  Patient 8 | 6
  Patient 9 | 7
  Patient 10 | 5
  Patient 11 | 7
  Patient 12 | 6
  Patient 13 | 6
  Patient 14 | 5
  Patient 15 | 6
  Patient 16 | 2
  Patient 17 | 4
  Patient 18 | 4
  Patient 19 | 4
  Patient 20 | 7
Percent Body Surface Area (BSA) Moveable Sclerosis at Baseline [Number; unit: Percent BSA moveable sclerosis] — Moveable sclerosis is also known as Morphea-like skin. Skin thickening that is full thickness and/or fixed to underlying bone and fascia.
  Percent BSA moveable sclerosis
    Patient 1 | 57.15
    Patient 2 | 2.7
    Patient 3 | 6.3
    Patient 4 | 0.18
    Patient 5 | 8.1
    Patient 6 | 59.4
    Patient 7 | 29.7
    Patient 8 | 15.3
    Patient 9 | 3.33
    Patient 10 | 0
    Patient 11 | 82.08
    Patient 12 | 12.6
    Patient 13 | 1.8
    Patient 14 | 5.4
    Patient 15 | 49.77
    Patient 16 | 0
    Patient 17 | 84.24
    Patient 18 | 15.84
    Patient 19 | 9.45
    Patient 20 | 0
Percent Body Surface Area (BSA) Nonmoveable Sclerosis at Baseline [Number; unit: Percent BSA nonmoveable sclerosis] — Non-moveable sclerosis is also known as non-hidebound thickened skin. Skin thickening that is full thickness and/or fixed to underlying bone and fascia.
  Percent BSA nonmoveable sclerosis
    Patient 1 | 7.56
    Patient 2 | 56.7
    Patient 3 | 36.9
    Patient 4 | 19.98
    Patient 5 | 77.94
    Patient 6 | 0
    Patient 7 | 32.4
    Patient 8 | 36.9
    Patient 9 | 9
    Patient 10 | 8.28
    Patient 11 | 0
    Patient 12 | 8.64
    Patient 13 | 71.1
    Patient 14 | 31.5
    Patient 15 | 10.8
    Patient 16 | 9.54
    Patient 17 | 0
    Patient 18 | 4.5
    Patient 19 | 11.7
    Patient 20 | 23.4
Baseline Range of Motion (ROM) Percent (of Predicted) [Number; unit: ROM Percent of Predicted] — This table lists the percentage of ROM present at baseline compared to expected ROM at a given joint. No measure of dispersion was performed because this is baseline data.
  ROM Percent of Predicted
    Patient 1 | 37
    Patient 2 | 56
    Patient 3 | 73
    Patient 4 | 7
    Patient 5 | 34
    Patient 6 | 47
    Patient 7 | 61
    Patient 8 | 35
    Patient 9 | 42
    Patient 10 | -7
    Patient 11 | 56
    Patient 12 | 37
    Patient 13 | 27
    Patient 14 | 32
    Patient 15 | 22
    Patient 16 | 71
    Patient 17 | 64
    Patient 18 | 54
    Patient 19 | 33
    Patient 20 | -5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Absolute Range of Motion (ROM) From Baseline to 6 Months
Description: A change in ROM is 25% or greater from baseline. A partial response required improvement in 25% or more in ROM. Progression required 25% or greater loss of ROM.Patients with negative values in the Table are those who lost ROM. Percent improvement in ROM for 1-3 target joints. For patients with >1 target joint, the average ROM improvement was calculated. The average percentage change in ROM deficit from baseline to 6 months was obtained based on the number of degrees of ROM change (6 months)/total ROM deficit (baseline) at each joint.
Time Frame: 6 months
Measure: Number; unit: Percent change from baseline
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 14
Percent change from baseline
  Pt 2 6mo response% change in deficit from baseline | 94
  Pt 7 6mo response% change in deficit from baseline | 35
  Pt 8 6mo response% change in deficit from baseline | 16
  Pt10 6mo response% change in deficit from baseline | 21
  Pt12 6mo response% change in deficit from baseline | 16
  Pt13 6mo response% change in deficit from baseline | 61
  Pt14 6mo response% change in deficit from baseline | 27
  Pt15 6mo response% change in deficit from baseline | 22
  Pt16 6mo response% change in deficit from baseline | 3
  Pt17 6mo response% change in deficit from baseline | -25
  Pt18 6mo response% change in deficit from baseline | -2
  Pt19 6mo response% change in deficit from baseline | 31
  Pt20 6mo response% change in deficit from baseline | 15

2. Primary Outcome: Primary Range of Motion (ROM) Response
Description: Progressive disease is defined as joint ROM: decrease of >25% in composite ROM score on 2 consecutive evaluations at least 2 weeks apart, but not greater than 4 weeks apart or steroid pulse: >1 steroid pulse per 3 month period if administered for sclerotic-type chronic graft versus host disease (ScGVHD). Response is joint ROM: increase of >25% in composite ROM score. Maximal response is a response with no further improvement over 2 sequential 3-month evaluations. Stable disease does not meet the criteria for progression, response, or maximal response.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 14
participants
  Partial Response | 5
  Stable Disease | 7
  Progressive Disease | 2

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately, 41 months, 27 days
Measure: Number; unit: Participants
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 20
Participants | 20

4. Secondary Outcome: Average Percentage Change in Range of Motion (ROM) Deficit
Description: One or more joints were assessed for ROM deficit by a physiatrist with expertise in graft versus host disease and joint ROM.
Time Frame: 6 months
Population: This outcome is the average percentage change in ROM deficit among 13 evaluable patients based on each patients baseline range of motion deficit compared to his/her ROM deficit at 6 months.
Measure: Mean (Inter-Quartile Range); unit: Percent change
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 13
Percent change | 24.2 [15.5 to 30.5]
Statistical Analysis 1: Comparison: Imatinib Mesylate in Patients With cGVHD; Test type: Superiority or Other; p = .011, Paired t-test

5. Secondary Outcome: Total Skin Score at Baseline and 6 Months
Description: Total skin score was graded by the National Institutes of Health Consensus Criteria. Skin score was calculated by dividing the total score by seven domains (skin, eye, oral, joint, gastrointestinal, hepatic, pulmonary) in men and 8 domains in women (previous domains noted plus gynecologic). Total skin score is a percentage of body surface area (BSA) involvement (range 0-100%). It was calculated from the sum of moveable body surface BSA and non-moveable BSA. Higher numbers = greater body surface area affected.
Time Frame: Baseline and 6 Months
Measure: Number; unit: units on a scale
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 14
units on a scale
  Patient # 2 - Baseline | 66.6
  Patient # 2 - 6 months | 54
  Patient # 3 - Baseline | 43.38
  Patient # 3 - 6 months | NA — This patient had progressive disease and was taken off study prior to 6 month endpoint. Hence, no data points at 6 months.
  Patient # 7 - Baseline | 66.24
  Patient # 7 - 6 months | 55.53
  Patient # 8 - Baseline | 53.1
  Patient # 8 - 6 months | 55.26
  Patient # 10 - Baseline | 10.8
  Patient # 10 - 6 months | 6.12
  Patient # 12 - Baseline | 21.24
  Patient # 12 - 6 months | 30.06
  Patient # 13 - Baseline | 79.2
  Patient # 13 - 6 months | 62.28
  Patient # 14 - Baseline | 39.96
  Patient # 14 - 6 months | 40.5
  Patient # 15 - Baseline | 71.46
  Patient # 15 - 6 months | 61.83
  Patient # 16 - Baseline | 9.54
  Patient # 16 - 6 months | 8.1
  Patient # 17 - Baseline | 84.96
  Patient # 17 - 6 months | 85.11
  Patient # 18 - Baseline | 26.64
  Patient # 18 - 6 months | 24.3
  Patient # 19 - Baseline | 21.15
  Patient # 19 - 6 months | 37.8
  Patient # 20 - Baseline | 23.4
  Patient # 20 - 6 months | 25.2

6. Secondary Outcome: Total Chronic Graft Versus Host Disease (cGVHD) Provider Global Rating Score at Baseline and 6 Months
Description: The provider global rating is a physician impression of severity of cGVHD symptoms from a scale of zero (no symptoms) to 10 (most severe GVHD symptoms possible).
Time Frame: Baseline and 6 months
Measure: Number; unit: Provider Global Rating Score
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 14
Provider Global Rating Score
  Patient #2 at Baseline | 5
  Patient #2 at 6 Months | 4
  Patient #3 at Baseline | 3
  Patient #3 at 6 Months | NA — This patient had progressive disease and was taken off study prior to 6 month endpoint. Hence, no data points at 6 months.
  Patient #7 at Baseline | 6
  Patient #7 at 6 Months | 8
  Patient #8 at Baseline | 6
  Patient #8 at 6 Months | 7
  Patient #10 at Baseline | 5
  Patient #10 at 6 Months | 4
  Patient #12 at Baseline | 6
  Patient #12 at 6 Months | 7
  Patient #13 at Baseline | 6
  Patient #13 at 6 Months | 4
  Patient #14 at Baseline | 7
  Patient #14 at 6 Months | 6
  Patient # 15 at Baseline | 7
  Patient #15 at 6 Months | 6
  Patient #16 at Baseline | 5
  Patient #16 at 6 Months | 4
  Patient #17 at Baseline | 6
  Patient #17 at 6 months | 8
  Patient #18 at Baseline | 8
  Patient #18 at 6 Months | 8
  Patient #19 at Baseline | 8
  Patient #19 at 6 Months | 5
  Patient #20 at Baseline | 8
  Patient #20 at 6 Months | 8
Statistical Analysis 1: Comparison: Imatinib Mesylate in Patients With cGVHD; Test type: Superiority or Other; p = .47, t-test, 2 sided

7. Secondary Outcome: Lung Function Score at Baseline and 6 Months
Description: Lung function was graded by the National Institutes of Health Chronic Graft Versus Host Disease organ response criteria. The Lung function score = forced expiratory volume 1 (FEV1) score + carbon monoxide diffusing capacity (DLCO) score, with a possible range of 2 (better outcome)-12 (worst outcome). The percent predicted FEV1 and DLCO (adjusted for hematocrit but not alveolar volume) should be converted to a numeric score as follows: >80% =1; 70-79% = 2; 60-69% = 3; 50-59% = 4; 40-49% = 5; <40% = 6.
Time Frame: Baseline and 6 Months
Measure: Number; unit: units on a scale
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 14
units on a scale
  Patient #2 at Baseline | 2
  Patient #2 at 6 Months | 2
  Patient #3 at Baseline | 9
  Patient #3 at 6 Months | NA — This patient had progressive disease and was taken off study prior to 6 month endpoint. Hence, no data points at 6 months.
  Patient #7 at Baseline | 3
  Patient #7 at 6 Months | 8
  Patient #8 at Baseline | 5
  Patient #8 at 6 Months | 6
  Patient #10 at Baseline | 3
  Patient #10 at 6 Months | 3
  Patient #12 at Baseline | 4
  Patient #12 at 6 Months | 5
  Patient #13 at Baseline | 4
  Patient #13 at 6 Months | 4
  Patient #14 at Baseline | 5
  Patient #14 at 6 Months | 5
  Patient # 15 at Baseline | 7
  Patient #15 at 6 Months | 6
  Patient #16 at Baseline | 3
  Patient #16 at 6 Months | 2
  Patient #17 at Baseline | 5
  Patient #17 at 6 months | 6
  Patient #18 at Baseline | 8
  Patient #18 at 6 Months | 8
  Patient #19 at Baseline | 9
  Patient #19 at 6 Months | 9
  Patient #20 at Baseline | 2
  Patient #20 at 6 Months | 2
Statistical Analysis 1: Comparison: Imatinib Mesylate in Patients With cGVHD; Test type: Superiority or Other; p = .29, t-test, 2 sided

8. Secondary Outcome: Change in Immunosuppression
Description: Change in immunosuppression was defined by an increase or decrease in steroid use form baseline.
Time Frame: 6 months
Population: Pred:prednisone; tacro:tacrolimus; MPred:methylprednisolone; siro:sirolimus; and MMF:mycophenolate mofetil
Measure: Number; unit: participants
Arm/Group | Imatinib Mesylate in Patients With cGVHD
Number analyzed (Participants) | 14
participants
  ↓ Pred 20 mg everyday (qd )to 5 mg every other day | 1
  ↓ MPred 16 mg every other day(qod) to 4 mg qod | 1
  ↓ Pred:24mg every day(qd) to 20mg qd | 1
  No change | 5
  ↓ Tacro 2mg every am 1.5mg every pm to .5mg bid | 1
  Pred↓ 25mg qd to 15mg qd;Tacro↓ 2mg bid to 1mg bid | 1
  Pred↓ 2.5mg qd to 2.5mg every other day | 1
  ↓ Siro:2mg qd to 1 mg qd | 1
  Pred wean then ↑ 10 12.5mg bid;Tacro↑1.0 to 1.5bid | 1
  MMF↓ 1g/bid to discontinued | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately, 41 months, 27 days.
Arm/Group | Imatinib Mesylate in Patients With cGVHD
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate in Patients With cGVHD (N=20)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema::head and neck (General disorders) | 1 (1)
Edema: limb (General disorders) | 1 (1)
Edema:: trunk/genital (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, Pulmonary edema) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate in Patients With cGVHD (N=20)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4 (8)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 5 (10)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (6)
Alkaline phosphatase (Investigations) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1)
CPK (creatine phosphokinase) (Investigations) | 5 (11)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Constitutional Symptoms-Other (Specify, cold intolerance; sleep walking) (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Creatinine (Investigations) | 2 (8)
Dermatology/Skin-Other (Specify, intermt. bilateral hands & L. hip) (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (19)
Dizziness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema::head and neck (General disorders) | 3 (6)
Edema: limb (General disorders) | 3 (11)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (22)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2)
Flu-like symptoms (General disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (2)
Glucose, serum-low (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (2)
Hemoglobin (Investigations) | 6 (13)
Hypertension (Vascular disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::otitis externa (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 1 (2)
leukoencephalopathy (radiographic findings) (Nervous system disorders) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (3)
Mood alteration::Depression (Psychiatric disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft tissue - Other (Specify, hand & jaw cramps; hand & jaw cramps, intermittent (Musculoskeletal and connective tissue disorders) | 1 (2)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (30)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain::Breast (Reproductive system and breast disorders) | 1 (1)
Pain::External ear (Ear and labyrinth disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 5 (11)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 6 (14)
Pain::Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 11 (26)
Platelets (Investigations) | 1 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (5)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (4)
Tinnitus (Ear and labyrinth disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-04-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT00702689/Prot_SAP_000.pdf
  • Informed Consent Form (2012-01-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT00702689/ICF_001.pdf